CLINICAL TRIAL: NCT05383495
Title: Anxiolysis for Laceration Repair in Children: A Multicenter Adaptive Randomized Trial
Brief Title: Anxiolysis for Laceration Repair in Children
Acronym: ALICE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DFS05081977
Record Dates: First submitted 2022-05-10; First posted 2022-05-20 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-03

CONDITIONS: Laceration of Skin; Distress, Emotional
MeSH Terms: interventions — Dexmedetomidine; Midazolam; Nitrous Oxide; Entonox

STUDY DESIGN:
Intervention Model Description: Phase III, multicentre, open-label, randomized, three-arm, adaptive trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intranasal dexmedetomidine (Experimental): IN dexmedetomidine 3 mcg/kg [100 mcg/mL (max 200 mcg or 2 mL)]
  Interventions: Drug: Dexmedetomidine
- Intranasal midazolam (Experimental): IN midazolam 0.4 mg/kg [5 mg/mL (max 10 mg or 2 mL)]
  Interventions: Drug: Midazolam Nasal Spray
- Inhaled nitrous oxide (Experimental): 50% N2O in 50% oxygen by face mask or on-demand system
  Interventions: Drug: Nitrous oxide

INTERVENTIONS:
Drug: Dexmedetomidine — Intranasal dexmedetomidine 3 mcg/kg [100 mcg/mL (max 200 mcg or 2 mL)
  Other Names: Precedex
  Arms: Intranasal dexmedetomidine
Drug: Midazolam Nasal Spray — Intranasal midazolam 0.4 mg/kg [5 mg/mL (max 10 mg or 2 mL)
  Other Names: Versed
  Arms: Intranasal midazolam
Drug: Nitrous oxide — 50% nitrous oxide in 50% oxygen by face mask
  Other Names: Nitronox
  Arms: Inhaled nitrous oxide

SUMMARY:
This is a 3-arm adaptive clinical trial to the optimal light sedative for reducing distress during laceration repair in children. The investigators will compare intranasal (IN) dexmedetomidine, IN midazolam, and nitrous oxide (N20). The primary outcome is the Observational Scale of Behavioral Distress - Revised (OSBD-R).

DETAILED DESCRIPTION:
Accounting for almost half of all procedures performed, lacerations are the most common reason for an ED visit in children. There is consistent evidence that children experience considerable distress during laceration repair, despite routine application of topical anesthetic, lidocaine-epinephrine-tetracaine (LET). Certified child life specialists (CCLSs) can help children cope with distress but are not widely available. Untreated distress in childhood can lead to anxiety, needle phobia, and fear of medical care as adults. The American Academy of Pediatrics and American Academy of Pediatric Dentistry strongly recommend minimizing discomfort and controlling behavior and movement during procedures but there is no specific guidance on laceration repair. Many children require pharmacologic anxiolysis for laceration repair but evidence for the most effective agent is lacking. Although anxiolytics such as midazolam and nitrous oxide (N2O) are frequently used, there are drawbacks including variable efficacy and nasal irritation in the case of midazolam and lack of cooperation in younger children in the case of N2O. IN dexmedetomidine is a potentially effective anxiolytic for laceration repair that could overcome these limitations.

IN dexmedetomidine is a relatively new anxiolytic with sedative and analgesic properties. It is tasteless, non-irritative, and highly concentrated (100 mcg/mL). A maximum dose of 200 mcg/2 mL can be given with 2 pairs of 0.5 mL IN sprays. The investigator's team published a systematic review of IN dexmedetomidine for distressing procedures. It was well tolerated by more than 90% of children and provided adequate anxiolysis in more children (79%) versus conventional anxiolytics (midazolam, chloral hydrate) (60%). Only one trial investigated IN dexmedetomidine in children for laceration repair and 70% were deemed "not anxious" compared to IN midazolam (11%). However, the study focused on initial positioning rather than repair. For proof of concept and to identify the optimal dose and feasibility of IN dexmedetomidine, we completed a pilot of 55 children undergoing laceration repair. All children tolerated IN administration, the consent rate was 82%, and there were no serious adverse events (AE). A dose of 3 mcg/kg balanced efficacy with duration of sedation, in line with others' findings.

Oral midazolam is the most common anxiolytic for laceration repair in children. However, onset and duration of action and efficacy can be unreliable and its bitter taste leads to poor compliance. IN midazolam using a mucosal atomizer device (MAD) is increasingly popular because it overcomes these limitations. Compared to oral midazolam, IN midazolam has a shorter onset of action (28 vs 34 minutes) but causes nasal irritation in up to 40% of patients. In addition, IN midazolam has variable efficacy for laceration repair and more adverse effects compared to nitrous oxide or IN dexmedetomidine. The largest study of IN midazolam was a retrospective study of combination IN midazolam plus fentanyl. A lower dose of midazolam (0.2 mg/kg) resulted in fewer adverse effects (0.7%) than with higher doses (2-5%). Adding IN fentanyl provided superior efficacy where only 2.4% of patients experienced a treatment failure.

The second most common anxiolytic is inhaled N2O, a tasteless gas that is administered in a concentration of 30-70% with oxygen. N2O is safe and effective for minor painful procedures. Peak effect is rapid (2 minutes) and effects dissipate quickly (3 minutes) upon discontinuation. Minor adverse effects occur in less than 10% of patients. However, based on the United Kingdom National Clinical Guideline Centre, it's unclear whether uncooperative children will comply with N2O administration. The investigators' recently completed systematic review of 29 trials of N2O for painful procedures in children found 50% N2O was superior to subcutaneous lidocaine, placebo, and oral midazolam. Only 5 trials focused on laceration repair but they were small and limited by non-validated or no measures of anxiety .

Despite frequent use of anxiolytics such as midazolam and N2O, The investigators' national survey found that 80% of Canadian paediatric ED physicians strongly believed that "children experience significant enough distress to warrant anxiolysis" and it would "improve the patient care experience". To improve care, a rigorous trial of a novel anxiolytic, IN dexmedetomidine, and dissemination of the research findings is needed.

ELIGIBILITY:
Inclusion Criteria:

i) Age 2-12.99 years [highest incidence of laceration repair] ii) Single or grouped lacerations separated by no more than 2 cm for which the treating physician believes repair does not require IV sedation iii) Repair to involve sutures and performed by ED physician or designate (trainee) iv) Child or caregiver desires anxiolysis for laceration repair [justification: incorporates family preferences based on their prior experiences or beliefs about child's response] vii) Local anesthesia planned to involve topical anesthetic (LET), infiltrated lidocaine, ring, or thenar block

Exclusion Criteria:

i) Sedative, anxiolytic, or alpha-2-adrenergic receptor agonist < 24 hours prior to interventions (may compound sedative effect and increase the SAE risk). 24-hours encompasses the duration of sedation of most agents.

ii) Hypersensitivity to any intervention iii) Occlusion of > 1 nostril due to polyps, septal deviation, or foreign body (may prevent drug absorption) iv) Hemodynamic abnormalities: bradycardia or hypotension < 2 SD of age-related normal value v) IND contraindications: Pre-existing renal insufficiency, uncorrected mineralocorticoid deficiency, pulmonary hypertension, uncorrected cyanotic heart disease, cardiac conduction disorder, pulmonary hypertension, pulmonary edema, vitamin B12 or folate disorder, phenylketonuria, or psychosis vi) Sedation contraindications: Impaired level of consciousness or respiratory instability vii) N2O contraindications: Conditions associated with potential accumulation of gas within body spaces viii) Suspected or confirmed pregnancy (as reported by patient) ix) Inability to vocalize pain due to motor deficits (unable to apply the OSBD-R) x) Caregiver unable to complete study tasks due to insufficient comprehension of either English or French in the absence of a native language interpreter xi) Weight >= 65 kg (to avoid under-dosing of INM or IND) x) Not American Society of Anesthesiologists class I (healthy) or II (controlled mild to moderate disease) xii) No concomitant fracture or dislocation requiring orthopedic manipulation

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Observational Scale of Behavioral Distress - Revised (OSBD-R) | During preparation, suturing, and recovery (20 minutes)
  Score ranges from 0 (no distress) to 23.5 (maximal distress) and will be scored for the time interval encompassing preparation and suturing

SECONDARY OUTCOMES:
Adverse effects | From intervention to 72 hours post-discharge
  Will be based on the Quebec Guidelines and Health Canada reporting standards for sedation in children and include nausea and vomiting
Need for additional anxiolysis or sedation to facilitate repair | During suturing (10 minutes)
  Need for additional anxiolysis or sedation to facilitate repair
Need for physical restraint | During preparation and suturing (10 minutes)
  Need for restraint during preparation and suturing based on the Procedural Restraint Intensity in Children (PRIC) scale. The PRIC is scored in discrete integer values from 0=no restraint to 4=extreme forceful restraint. A higher score indicates more restraint is needed.
Late maladaptive behaviors | From discharge to 72 hours post-discharge
  Late maladaptive behaviors up to an including 72 hours post discharge using the Post-Hospital Behavior Questionnaire. The scale consists of 27 items concerning sleep, eating, anxiety, etc. where each item is scored from 1-5. The minimum score is 27 and the maximum score is 135 with higher scores indicating greater severity of behaviors.

OTHER OUTCOMES:
Compliance with intervention administration | From drug administration through completion of suturing (40 minutes)
  Compliance (percent of calculated IN volume given and acceptance of face mask or on-demand mouthpiece (yes/no))
Caregiver satisfaction with anxiolysis during laceration repair | At discharge (1 minute)
  Caregiver satisfaction with anxiolysis using a 100 mm visual analog scale. A higher score indicates greater satisfaction.
Child satisfaction with anxiolysis during laceration repair | At discharge (1 minute)
  Child (7-12 years) satisfaction with anxiolysis using a 100 mm visual analog scale. A higher score indicates greater satisfaction.
Healthcare provider (physician, nurse, respiratory therapist) satisfaction with anxiolysis during laceration repair | During recovery (1 minute)
  Nurse, physician, parent, and child 7-12 years satisfaction with anxiolysis using a 100 mm visual analog scale. A higher score indicates greater satisfaction.
Number of healthcare personnel required during repair | During procedure (10 minutes)
  Maximum number of healthcare personnel required at bedside during repair to provide physical restraint or patient care
Cost of healthcare personnel required at bedside during repair | During procedure (40 minutes)
  Costs of healthcare personnel based on salary per minute required at bedside during repair to provide physical restraint or patient care
Cost of interventions | During procedure (40 minutes)
  Cost of interventions based on group assignment
Total ED length of stay | During emergency department visit (2 hours)
  ED length of stay
Duration of procedure | During procedure (40 minutes)
  Duration of laceration repair
Post-intervention length of stay | From drug administration to discharge (80 minutes)
  Length of stay due to anxiolytic
Nasal irritation | During IN intervention administration (2 minutes)
  Nasal irritation due IN intervention using the FLACC scale. Measured following IN sprays
Post-procedure length of stay | From suturing to discharge (40 minutes)
  Post-procedure length of stay
Caregiver state anxiety | Immediately prior to Phase II (preparation) (1 minute)
  Caregiver anxiety related to laceration repair using State Trait Anxiety Inventory Short version - State (STAIS5)

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jiang A, Poonai N, Arthur-Hayward V, Heath A. Anxiolysis for laceration repair in children: statistical analysis plan for an open-label multicenter adaptive trial (ALICE). Trials. 2025 Aug 7;26(1):280. doi: 10.1186/s13063-025-09009-z. PMID 40775649
- [Derived] Poonai N, Arthur-Hayward V, Ali S, Sabhaney V, Doan Q, Trottier E, Gravel J, Tran NA, Bhatt M, Eltorki M, Thull-Freedman J, Leung J, Beer D, Jiang A, Poolacherla R, Heath A. Anxiolysis for laceration repair in children: study protocol for an open-label multicenter adaptive trial (ALICE). PLoS One. 2025 Jun 4;20(6):e0324515. doi: 10.1371/journal.pone.0324515. eCollection 2025. PMID 40465577